CLINICAL TRIAL: NCT03747783
Title: Development and Validation of Nomograms to Precisely Predict Conditional Risk of Survival for Patients With Laryngeal Cancer: a Single-institutional Study
Brief Title: Nomograms to Precisely Predict Conditional Risk of Survival for Patients With Laryngeal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, GengLong Liu, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: Laryngeal cacer
Record Dates: First submitted 2018-11-17; First posted 2018-11-20 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Laryngeal Cancer
Keywords: Survival; Nomograms; Laryngeal cancer
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survival Group: status from radical operation to follow-up
  Interventions: Procedure: Radical Operation
- Non-Survival Group: status from radical operation to follow-up
  Interventions: Procedure: Radical Operation

INTERVENTIONS:
Procedure: Radical Operation — The surgery treatment selection was based on the American Joint Committee on Cancer stage both of the primary and of the recurrence, as well as on patterns of local spread that were not included in the T classification and on the general condition and preferences of each patient.

SUMMARY:
Advanced laryngeal squamous cell carcinoma (SCC) remains a highly morbid and fatal disease despite aggressive interventions. Mortality is high in this cohort: laryngeal cancer affects over 13 000 patients in the United States, with over 3500 deaths annually.The results of the Veterans Affairs Cooperative Studies Program Laryngeal Cancer Trial and subsequent studies demonstrated similar overall survival (OS) rates for organ preservation protocols involving radiotherapy (RT) or chemoradiotherapy (CRT) when compared to surgery, with the benefit of preserving the larynx in a large majority of patients. As such, the use of RT or CRT has become the predominant initial intervention for patients with laryngeal SCC.However, the prognosis of recurrent and persistent laryngeal SCC is particularly dire.In this study,the investigators sought to identify preoperative predictors of survival for patients with recurrent or persistent laryngeal SCC in order to set patient expectations and address modifiable risk factors. Identification of predictors of survival may also identify patients who could benefit from novel therapeutic agents in a neo/adjuvant fashion. Herein,we examine a cohort of patients with recurrent or persistent laryngeal SCC after definitive RT/CRT who has undergone total laryngectomy in order to identify potential preoperative predictors of clinical outcomes.

DETAILED DESCRIPTION:
Demographic, clinical, and survival data were abstracted. Death was verified via medical records and the social security death index. Primary outcome measures were OS (time from salvage laryngectomy to death from any cause), disease-specific survival (DSS; time from salvage laryngectomy to death from recurrent/persistent laryngeal SCC), and DFS (time from salvage laryngectomy to laryngeal SCC recurrence)

ELIGIBILITY:
Inclusion Criteria:

* laryngeal carcinoma patients with radical surgery

Exclusion Criteria:

* multiple primarry malignant neo-plasms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: laryngeal carcinoma patients with radical surgery
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-01-03 (Actual); Primary Completion 2019-01-03 (Estimated); Study Completion 2019-03-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Follow up 5 year
  time from laryngectomy to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Tan, Study Chair — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (1):
- Genglong Liu, Guangzhou, State..., China

IPD SHARING:
Plan to Share IPD: Undecided